CLINICAL TRIAL: NCT03467152
Title: A Placebo-Controlled, Double-Blind, Parallel-Group, Randomized, Study To Evaluate the Efficacy, Safety and Tolerability of E2027 in Subjects With Dementia With Lewy Bodies
Brief Title: Study To Evaluate the Efficacy, Safety and Tolerability of E2027 (Hereinafter Referred to as Irsenontrine) in Participants With Dementia With Lewy Bodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2027-G000-201; 2017-003728-64 (EudraCT Number)
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Dementia With Lewy Bodies
Keywords: Irsenontrine; Montreal Cognitive Assessment; Neuropsychiatric Inventory; Mini-Mental State Examination; Cognitive Fluctuation Inventory
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Irsenontrine (Experimental): Participants will be randomized to receive a 50 milligram (mg) once daily oral dose of Irsenontrine for 12 weeks.
  Interventions: Drug: Irsenontrine
- Placebo (Placebo Comparator): Participants will be randomized to receive a 50 mg once daily oral dose of Irsenontrine-matched placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irsenontrine — Oral hypromellose capsules.
  Other Names: E2027
  Arms: Irsenontrine
Drug: Placebo — Oral hypromellose capsules.
  Arms: Placebo

SUMMARY:
This study will be conducted to compare Irsenontrine to placebo on the cognitive endpoint of Montreal Cognitive Assessment (MoCA) and the global clinical endpoint of Clinician's Interview Based Impression of Change Plus (CIBIC-Plus) Caregiver Input in participants with dementia with Lewy bodies after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 50 to 85 years, inclusive at time of consent.
* Meet criteria for probable dementia with Lewy bodies (DLB) (as defined by the 4th report of the DLB Consortium).
* Mini-Mental State Examination greater than or equal to (≥)14 and less than or equal to (≤) 26 at Screening Visit.
* Has experienced visual hallucinations during the past 4 weeks before Screening Visit.
* If receiving acetylcholinesterase inhibitors (AChEI), must have been on a stable dose for at least 12 weeks before Screening Visit, with no plans for dose adjustment during the study. Treatment-naive participants can be entered into the study but there should be no plans to initiate treatment with AChEIs from Screening to the end of the study.
* If receiving memantine, must have been on a stable dose for at least 12 weeks before Screening Visit, with no plans for dose adjustment during the study. Treatment naive participants can be entered into the study but there should be no plans to initiate treatment with memantine from Screening to the end of the study.
* Must have an identified caregiver or informant who is willing and able to provide follow-up information on the participant throughout the course of the study.
* Provide written informed consent. If a participant lacks capacity to consent in the investigator's opinion, the participant's assent should be obtained, as required in accordance with local laws, regulations and customs, plus the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations). In countries where local laws, regulations, and customs do not permit participants who lack capacity to consent to participate in this study, they will not be enrolled.

Exclusion Criteria:

* Any neurological condition that may be contributing to cognitive impairment above and beyond those caused by the participant's DLB, including any comorbidities detected by clinical assessment or magnetic resonance imaging (MRI).
* History of transient ischemic attacks or stroke within 12 months of Screening.
* Modified Hachinski Ischemic Scale greater than (>) 4.
* Parkinsonian (extrapyramidal) features with Hoehn and Yahr stage 4 intravenous or higher.
* Any major psychiatric diagnosis, including schizophrenia, bipolar disorder and current major depressive disorder as per Diagnostic and Statistical Manual of Mental Disorders Fifth Edition.
* Geriatric Depression Scale score > 8.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (25):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - Parkinsons and Movement Disorders Institute, Fountain Valley, California
  - Paradigm Clinical Research Centers, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Miami Jewish Health-Clinical Research, Miami, Florida
  - Elias Research Associates (Allied Biomedical Research Institute), Miami, Florida
  - Pharmax Research of South Florida; Elias Research Associates, Miami, Florida
  - Compass Research-Bioclinica, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Compass Research-Bioclinica, The Villages, Florida
  - Indiana University, Dept of Neurology, Indianapolis, Indiana
  - University of Kentucky, Dept of Neurology Sanders Brown Center on Aging, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Neurological Associates of Albany, PC, Albany, New York
  - Columbia University, New York, New York
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Cleveland Clinic, Lou Ruvo Center for Brain Health at Lakewood Hospital, Lakewood, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Kerwin Research Center, LLC, Dallas, Texas
  - University of Virginia Adult Neurology, Charlottesville, Virginia
- France (6):
  - CHRU Nancy- CMRR de lorraine Hôpital de Brabois-Service de Gériatrie, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre de Recherche Clinique - Viellissement-Cerveau-Fragilite (CRC-VCF), Hopital des Charpennes, Lyon, Villeurbanne
  - Centre Memoire du CHRU de Lille, Lille
  - Hopital Neurologique de Lyon, Lyon
  - University Hospital de la Timone, Marseille
  - Centre d'Investigation Clinique (CIC) Hopitaux universitaires Strasbourg HOPITAL DE HAUTEPIERRE - BATIMENT AX5, Strasbourg
- Germany (3):
  - Eisai Trial Site #3, Berlin
  - Eisai Trial Site #1, Kassel
  - Eisai Trial Site #2, Westerstede
- Italy (2):
  - Universita Chieti, CeSI Met, Chieti
  - Clinica Neurologica Azienda Ospedaliera di Padova, Padua
- Japan (23):
  - Eisai Trial Site #20, Chiba, Chiba
  - Eisai Trial Site #17, Fukuoka, Fukuoka
  - Eisai Trial Site #8, Fujioka-shi, Gunma
  - Eisai Trial Site #12, Maebashi, Gunma
  - Eisai Trial Site #14, Miyoshi-shi, Hiroshima
  - Eisai Trial Site #4, Otake-shi, Hiroshima
  - Eisai Trial Site #2, Himeji-shi, Hyōgo
  - Eisai Trial Site #23, Yokohama, Kanagawa
  - Eisai Trial Site #11, Kumamoto, Kumamoto
  - Eisai Trial Site #5, Nishisonogigun, Nagasaki
  - Eisai Trial Site #9, Nagaoka-shi, Niigata
  - Eisai Trial Site #3, Kurashiki-shi, Okayama-ken
  - Eisai Trial Site #1, Naniwa-ku, Osaka
  - Eisai Trial Site #16, Sakai-ku, Sakai-shi, Osaka
  - Eisai Trial Site #24, Suita-shi, Osaka
  - Eisai Trial Site #13, Suita-shi, Osaka
  - Eisai Trial Site #6, Kanzaki-gun, Saga-ken
  - Eisai Trial Site #10, Bunkyo-ku, Tokyo
  - Eisai Trial Site #22, Mitaka-shi, Tokyo
  - Eisai Trial Site #18, Setagaya-Ku, Tokyo
  - Eisai Trial Site #19, Yanai-shi, Yamaguchi
  - Eisai Trial Site #25, Hiroshima
  - Eisai Trial Site #21, Osaka
- Spain (6):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Institut Internacional de Neurociències Aplicades, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
- United Kingdom (9):
  - Dementia Research Unit, Crowborough, East Sussex
  - Memory Assessment and Research Centre, Moorgreen Hospital, Southampton, Hampshire
  - Clinical Research Centre (CRC), Dundee, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - West London Mental Health Trust, Isleworth
  - Kings College, London
  - Cognition Health, London
  - Manchester Mental Health and Social Care Trust, Manchester
  - Newcastle General Hospital, Newcastle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 investigative sites in the United States, Japan, United Kingdom, France, Spain, Germany, and Italy from 04 May 2018 to 15 April 2020.
Pre-assignment Details: A total of 326 participants were enrolled (signed informed consent form), of which 120 were screen failures and 206 were randomized, out of which 196 were treated. 6 participants were randomized at a site that was subsequently closed for serious compliance issues. The treatment arms to which these 6 participants were randomized is unknown and no data was collected for the Baseline, Outcome Measures, and Adverse Events module. These 6 participants were excluded from all analyses.
Groups:
- Placebo: Participants received Irsenontrine-matched placebo capsule, orally, once daily for 12 weeks.
- Irsenontrine 50 mg: Participants received Irsenontrine 50 milligram (mg), capsule, once daily for 12 weeks.
- Randomised, Not Treated Due to Site Closure: 6 participants were randomized at a site that was subsequently closed for serious compliance issues. The treatment arms to which these 6 participants were randomized is unknown and no data was collected for the Baseline, Outcome Measures, and Adverse Events module.
Period: Overall Study
Arm/Group | Placebo | Irsenontrine 50 mg | Randomised, Not Treated Due to Site Closure
Started | 100 | 100 | 6 (The treatment arms to which these 6 participants were randomized is unknown.)
Treated | 97 | 99 | 0
Completed | 84 | 89 | 0
Not Completed | 16 | 11 | 6
Not completed — Adverse Event | 4 | 5 | 0
Not completed — Subject Choice | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0
Not completed — Others | 3 | 0 | 0
Not completed — Not treated | 3 | 1 | 6

BASELINE CHARACTERISTICS:
Population: The safety analysis set included the group of participants who received at least 1 dose of study drug and had at least 1 post randomization safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Irsenontrine 50 mg | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.8 (6.60) | 75.3 (6.44) | 74.5 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 61 | 62 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 17 | 28
  Not Hispanic or Latino | 73 | 76 | 149
  Unknown or Not Reported | 13 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 34 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 48 | 55 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montreal Cognitive Assessment (MoCA) Total Score at Week 12 of Treatment
Description: The MoCA scale is used for detecting cognitive impairment. The scores range between 0 to 30 points; a score of 26 or above was considered normal. Higher values represent a better outcome.
Time Frame: Baseline and Week 12
Population: The full analysis set included the group of randomized participants who received at least 1 dose of study drug, had baseline and at least 1 post randomization coprimary efficacy measurement. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure and number analyzed "n" are the participants who were evaluable for the outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 92 | 96
score on a scale
  Baseline | 13.9 (5.40) | 13.8 (5.18)
  Change at Week 12: number analyzed (Participants) | 81 | 87
  Change at Week 12 | -0.6 (2.63) | -0.4 (3.41)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.6909, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

2. Primary Outcome: Number of Participants Based on Clinician's Interview Based Impression of Change Plus Caregiver Input (CIBIC-Plus) Scale at Week 12 of Treatment
Description: Number of participants are reported categorized in grades based on the CIBIC-Plus scale. The CIBIC-Plus scale is designed to measure various domains that describe participant function: general, mental/cognitive state, behavior, and activities of daily living. It is a semi-structured global rating derived from a comprehensive interview with the participant and caregiver or informant by an independent rater who has no access to the source data or other psychometric test scores conducted post-randomization as part of the protocol. The CIBIC-Plus was a 7-point scale and scores were: 1 (marked improvement), 2 (moderate improvement), 3 (minimal improvement), 4 (no change), 5 (minimal worsening), 6 (moderate worsening), and 7 (marked worsening). Higher values represent a worse outcome.
Time Frame: Week 12
Population: The full analysis set included the group of randomized participants who received at least 1 dose of study drug, had baseline and at least 1 post randomization coprimary efficacy measurement. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 86 | 89
Participants
  Marked improvement | 0 | 0
  Moderate improvement | 5 | 3
  Minimal improvement | 13 | 18
  No change | 32 | 32
  Minimal worsening | 30 | 28
  Moderate worsening | 6 | 8
  Marked worsening | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.8251, GLMM — Generalized Linear Mixed Models Analysis (GLMM); Odds Ratio (OR) = 1.018, 95% CI 2-sided [0.695 to 1.492]

3. Secondary Outcome: Clinician's Global Impression of Change - In Dementia With Lewy Bodies (CGIC-DLB) Scale at Week 12 of Treatment
Description: Number of participants are reported categorized in grades based on the CGIC-DLB scale. The CGIC-DLB scale provided an overall clinician-determined summary measure of change from the participant's clinical status that takes into account all available information from the efficacy endpoints (which include cognitive function, non-cognitive symptoms, behavior, and the impact of the symptoms on the participant's ability to function) and safety data. The (CGIC-DLB) was a 7-point scale and scores were: 1 (marked improvement), 2 (moderate improvement), 3 (minimal improvement), 4 (no change), 5 (minimal worsening), 6 (moderate worsening), and 7 (marked worsening). Higher values represent a worse outcome.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 83 | 90
Participants
  Marked improvement | 1 | 0
  Moderate improvement | 3 | 10
  Minimal improvement | 20 | 15
  No change | 36 | 30
  Minimal worsening | 22 | 27
  Moderate worsening | 1 | 8
  Marked worsening | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.3003, GLMM — Generalized Linear Mixed Models Analysis (GLMM); Odds Ratio (OR) = 0.853, 95% CI 2-sided [0.584 to 1.247]

4. Secondary Outcome: Mean Change From Baseline in the Cognitive Fluctuation Inventory (CFI) Score at Week 12 of Treatment
Description: The CFI scale assessed cognitive fluctuation. It evaluates fluctuation in various domains including attention, ability to perform daily functions, orientation, verbal communication and behavior. The score was based on frequency and severity with a score range of 0 to 12. The scale also assessed the degree of caregiver or informant distress engendered by the symptoms. Higher scores indicating greater impairment.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 92 | 96
score on a scale
  Baseline | 3.4 (2.68) | 3.1 (2.48)
  Change at Week 12: number analyzed (Participants) | 86 | 89
  Change at Week 12 | 0.1 (3.20) | 0.3 (3.25)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.9198, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

5. Secondary Outcome: Mean Change From Baseline in the Mini-Mental State Examination (MMSE) Total Score Week 12 of Treatment
Description: The MMSE is a 30-point scale that measured orientation to time and place, registration, immediate and delayed recall, attention, language, and drawing. The total score ranges from 0 (most impaired) to 30 (no impairment). The lower score means severe cognitive deficit and higher score indicates better function.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 93 | 96
score on a scale
  Baseline | 21.0 (3.63) | 21.1 (3.22)
  Change at Week 12: number analyzed (Participants) | 85 | 92
  Change at Week 12 | -1.1 (3.63) | -1.7 (3.58)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.2909, ANCOVA

6. Secondary Outcome: Mean Change From Baseline in the Neuropsychiatric Inventory (NPI-12) Total Score at Week 12 of Treatment
Description: The NPI-12 scale assessed the frequency and severity of 12 neuropsychiatric symptoms commonly described in dementia participants: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating changes. The scale also assessed the degree of caregiver or informant distress engendered by each of the symptoms. The sum of the composite scores for the 12 domains yielded the NPI-12 total score. NPI-12 total score ranged from 0 (minimum severity) to 144 (maximum severity); higher score indicates greater neuropsychiatric disturbance.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 93 | 96
score on a scale
  Baseline | 17.6 (14.32) | 19.1 (16.07)
  Change at Week 12: number analyzed (Participants) | 86 | 89
  Change at Week 12 | -0.2 (11.07) | -2.0 (15.36)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.6127, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

7. Secondary Outcome: Change From Baseline in NPI-4 Subscore at Week 12
Description: The NPI scale assesses the frequency and severity of 12 neuropsychiatric symptoms commonly described in dementia participants: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating changes. NPI-4 is the subscore covering the domains of delusions, hallucinations, apathy and depression. NPI-4 total subscore ranged from 0 to 48, with higher scores indicating a greater neuropsychiatric disturbance.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 93 | 96
score on a scale
  Baseline | 8.2 (6.40) | 8.6 (7.18)
  Change at Week 12: number analyzed (Participants) | 86 | 89
  Change at Week 12 | -0.4 (5.15) | -0.6 (6.79)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.8780, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

8. Secondary Outcome: Change From Baseline in NPI-10 Subscore at Week 12
Description: The NPI-10 assessed range of behaviors seen in dementia for both frequency and severity. It is a 10 item questionnaire with the following domains: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/liability and aberrant motor behavior. The total score was a sum of the 10 domains, where the score of each domain was calculated as frequency (scale: 1=occasionally to 4=very frequently)*Severity (scale: 1=Mild to 3=Severe). Each domain has a maximum score of 12 and all domains were equally weighted for total score, the range for total score is 0 to 120. Higher scores indicating a greater neuropsychiatric disturbance.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 93 | 96
score on a scale
  Baseline | 13.5 (11.22) | 14.9 (13.54)
  Change at Week 12: number analyzed (Participants) | 86 | 89
  Change at Week 12 | 0.6 (9.32) | -1.4 (12.53)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.4090, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

9. Secondary Outcome: Change From Baseline in NPI-D (Caregiver Distress) Total Score at Week 12
Description: The NPI-D scale assesses the frequency and severity of 12 neuropsychiatric symptoms commonly described in dementia participants: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating changes. The scale assesses the degree of caregiver distress engendered by each of the symptoms. The caregiver distress (NPI-D) is rated by caregiver based on his or her own stress on a five point scale from 0 to 5, where: 0(no distress), 1(minimal), 2(mild), 3(moderate), 4(moderately severe), 5(very severe or extreme). NPI-D total score is calculated by summing the scores of the 12 sub-scale distress scores. The NPI-D total scores ranges from 0 to 60 with higher scores indicating greater distress.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 93 | 96
score on a scale
  Baseline | 8.8 (7.65) | 9.4 (8.44)
  Change at Week 12: number analyzed (Participants) | 86 | 89
  Change at Week 12 | -0.2 (6.18) | -0.6 (7.28)
Statistical Analysis 1: Comparison: Placebo vs Irsenontrine 50 mg; Test type: Superiority; p = 0.8736, MMRM — Mixed Models for Repeated Measures Analysis (MMRM)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Severe TEAEs, Serious TEAEs, Adverse Events (AEs) Resulting in Study Discontinuation
Description: A TEAE was defined as an AE that emerged or worsened in severity relative to baseline during treatment or within 28 days after the last dose of study drug. Severe TEAE was defined as inability to work or to perform normal daily activity. A Serious TEAE is any untoward medical occurrence that at any dose: results in death; is life threatening (that is, the participant was at immediate risk of death from the adverse event as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death) requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria. An adverse event (AE) was defined as any untoward medical occurrence in a participant administered an investigational product.
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 97 | 99
Participants
  TEAEs | 67 | 70
  Severe TEAEs | 6 | 2
  Serious TEAEs | 9 | 7
  AE Leading to Discontinuation from Study | 7 | 6

11. Secondary Outcome: Number of Participants With Orthostatic Hypotension
Description: Orthostatic hypotension was defined as drop in standing systolic blood pressure greater than or equal to (>=) 20 Millimeter of mercury (mmHg) compared to supine, or drop in standing diastolic blood pressure >=10 mmHg compared to supine.
Time Frame: Week 2, Week 4, Week 6, Week 9 and Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 97 | 99
Participants
  Week 2 | 10 | 2
  Week 4 | 9 | 7
  Week 6 | 6 | 11
  Week 9 | 13 | 9
  Week 12 | 7 | 9

12. Secondary Outcome: Number of Participants With Orthostatic Tachycardia
Description: Orthostatic tachycardia by numerical criteria was defined by the following numerical criteria: Standing heart rate (HR) increased by >30 beats/min compared to supine and absolute standing HR was >100 beats/min.
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 97 | 99
Participants | 1 | 0

13. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: A laboratory value was determined to be a markedly abnormal value if the postbaseline common toxicity criteria grade increased from baseline and the post-baseline grade was greater than or equal to 2.
Time Frame: From first dose of study drug up to Week 16
Population: The safety analysis set included the group of participants who received at least 1 dose of study drug and had at least 1 post randomization safety assessment. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure. Number analyzed "n" are the participants who were evaluable for the outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 94 | 97
Participants
  Albumin: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Albumin: Markedly Abnormal Low | 1 | 0
  Bilirubin: Markedly Abnormal High: number analyzed (Participants) | 94 | 96
  Bilirubin: Markedly Abnormal High | 1 | 0
  Calcium: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Calcium: Markedly Abnormal Low | 1 | 0
  Creatinine: Markedly Abnormal High: number analyzed (Participants) | 94 | 96
  Creatinine: Markedly Abnormal High | 0 | 2
  Gamma Glutamyl Transferase: Markedly Abnormal High: number analyzed (Participants) | 94 | 96
  Gamma Glutamyl Transferase: Markedly Abnormal High | 2 | 0
  Hemoglobin: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Hemoglobin: Markedly Abnormal Low | 0 | 1
  Leukocytes: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Leukocytes: Markedly Abnormal Low | 0 | 1
  Lymphocytes: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Lymphocytes: Markedly Abnormal Low | 4 | 1
  Neutrophils: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Neutrophils: Markedly Abnormal Low | 1 | 1
  Phosphate: Markedly Abnormal Low: number analyzed (Participants) | 94 | 96
  Phosphate: Markedly Abnormal Low | 0 | 1
  Potassium: Markedly Abnormal Low | 1 | 0
  Potassium: Markedly Abnormal High | 2 | 0

14. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Time Frame: From first dose of study drug up to Week 16
Population: The safety analysis set included the group of participants who received at least 1 dose of study drug and had at least 1 post randomization safety assessment. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 96 | 98
Participants
  QTcF prolongation by >60 milliseconds (ms) from baseline and absolute QTcF >450 ms | 2 | 0
  QTcF prolongation to >500 ms | 2 | 0
  Change from baseline of PR >= 25 percent (%) to an absolute PR value of >220 msec | 1 | 1
  Change from baseline of QRS >= 25% to an absolute QRS value of >120 msec | 1 | 0

15. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories); is an interview-based instrument to systematically assess suicidal ideation and suicidal behavior. C-SSRS assess whether participant experience any of the following: completed suicide; suicide attempt (response of "yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). Here, number of participants with positive response ("yes") to suicidal behavior or/and Ideation, any non-suicidal self-injurious behavior was reported.
Time Frame: From first dose of study drug up to Week 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 95 | 98
Participants
  Completed Suicide | 0 | 0
  Suicide Attempt | 0 | 0
  Preparatory Actions Towards Imminent Suicidal Behavior | 0 | 2
  Wish to Die | 6 | 8
  Actual Suicidal Thoughts; Non-specific | 1 | 1
  Actual Suicidal Thoughts with Method; No Intent | 0 | 1
  Active Thoughts with Intent | 0 | 0
  Active Thoughts with Plan and Intent | 0 | 0
  Self-injurious Behavior; No Intent | 0 | 0

16. Secondary Outcome: Change From Baseline in Total Score of Unified Parkinson's Disease Rating Scale Part III: Motor Examination (UPDRS-III)
Description: The UPDRS scale evaluates extrapyramidal features in motor function in Parkinson's disease. It contains 33 items in 18 categories: (1) speech, (2) facial expression, (3) rigidity, (4) finger tapping, (5) hand movements, (6) supinational and pronation movements of hands, (7) toe tapping, (8) leg agility, (9) arising from chair, (10) gait, (11) freezing of gait, (12) postural stability, (13) posture, (14) body bradykinesia, (15) postural tremor of hands, (16) kinetic tremor of hands, (17) rest tremor amplitude and (18) constancy of rest tremor. Each item is scored 0 to 4, giving a total score range 0 to 132. Higher scores indicating more severe symptoms.
Time Frame: Baseline up to Week 16
Population: The safety analysis set included the group of participants who received at least 1 dose of study drug and had at least 1 post randomization safety assessment. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Irsenontrine 50 mg
Number analyzed (Participants) | 97 | 99
score on a scale
  Baseline | 31.3 (18.51) | 34.5 (18.12)
  Change at Week 16: number analyzed (Participants) | 81 | 84
  Change at Week 16 | -1.2 (10.97) | 1.0 (9.22)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to follow up (Week 16)
Arm/Group | Placebo | Irsenontrine 50 mg
All-Cause Mortality (participants affected / at risk) | 1/97 | 0/99
Serious Adverse Events (participants affected / at risk) | 9/97 | 7/99
Other Adverse Events (participants affected / at risk) | 65/97 | 68/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Irsenontrine 50 mg (N=99)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 1 (1) | 2 (2)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Irsenontrine 50 mg (N=99)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 15 (15) | 10 (14)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 2 (2)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Norovirus test positive (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 4 (4)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (4) | 5 (5)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 2 (2) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Visuospatial deficit (Nervous system disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 2 (3)
Confusional state (Psychiatric disorders) | 2 (2) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 9 (11) | 7 (8)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 2 (2) | 0 (0)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Sexually inappropriate behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03467152/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03467152/SAP_003.pdf